CLINICAL TRIAL: NCT00174681
Title: Testing the Usefulness of Lantus When Initiated Prematurely In Patients With Type 2 Diabetes
Brief Title: Tulip Study: Testing the Usefulness of Lantus When Initiated Prematurely In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4042
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine

SUMMARY:
Primary objective:

The primary objective of this trial is:

* To evaluate the efficacy of initiating Lantus in combination with oral antidiabetics drugs compared to oral antidiabetic treatment optimised by enhancing hygienic and dietary measures in type 2 diabetics whose blood glucose control is acceptable but not optimal on maximum oral treatment, based on the number of patients achieving a HbA1c value < 7% at the end of treatment.

Secondary objectives:

The secondary objectives of this trial are to compare between the two treatment groups:

* The variation in HbA1c between baseline and end of trial.
* The frequency of episodes of symptomatic hypoglycaemia (diurnal and nocturnal), severe hypoglycaemia (diurnal and nocturnal) and asymptomatic hypoglycaemia.
* Mean blood glucose levels at different times of the day.
* The variation in weight and lipid in each group between baseline and end of trial.
* The incidence of adverse events.

ELIGIBILITY:
Inclusion criteria :

Subjects fulfilling all of the following criteria will be eligible for inclusion in the trial:

* Type 2 diabetes
* 24 ≤ BMI ≤ 35 kg/m2
* 7 % ≤ HbA1c ≤ 8 %
* Treated with OAD for at least 2 years
* Treated with at least two oral antidiabetics including one sulphonylurea at the maximum tolerated dosages and metformin at the maximum tolerated dosages
* Not treated with a glinide or thiazolidinedione.
* Capable of performing blood glucose self-monitoring and a self-injection of insulin.
* Funduscopy within the previous year at the time of inclusion.

Exclusion Criteria:

Patient with any of the following criteria will not be included in the trial:

* Type 1 diabetics
* Insulin-treated type 2 diabetics or having previously received long-term insulin, or treated with a thiazolidinedione or glinide
* Fasting blood glucose < 1.20 g/l.
* Pregnancy (non-menopausal women must have a pregnancy test before the inclusion visit and effective contraception).
* Lactation.
* History of hypersensitivity to the investigational product or to drugs with similar chemical structures.
* Systemic treatment with corticosteroids irrespective of the dose and irrespective of the previous or anticipated duration of treatment.
* Treatment with another product under development in the 2 months preceding the date of inclusion in the study.
* Subject likely to receive treatments prohibited in the protocol during the trial.
* Cardiovascular, hepatic, neurological, endocrine or any other disease making it difficult to carry out the protocol or interpret the results.
* Proliferative or rapidly progressive or unstable retinopathy for at least 6 months after treatment by surgery or laser, or requiring surgery or laser in the 3 months following inclusion in the study.
* Hepatic impairment:ALT and/or AST more than three times the upper limit of normal at the initial assessment.
* Renal insufficiency:Serum creatinine >177 µmol/l (>20 mg/l) or creatinine clearance <60 ml/min.
* Previous or current history of alcohol or drug abuse.
* Mental state rendering the subject incapable of understanding the nature, objectives and possible consequences of the trial.
* Inability to undertake blood glucose self-monitoring and the injection of insulin alone.
* Subject unable to accept the restrictions of the protocol (uncooperative, unable to attend the follow-up visits and probably incapable of completing the trial).
* Subjects deprived of freedom by an administrative or judicial decision.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2003-04

PRIMARY OUTCOMES:
Percentage of subjects achieving HbA1c < 7% at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis, Zagreb, Croatia
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Bucharest, Romania
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Ljubljana, Slovenia